CLINICAL TRIAL: NCT05886062
Title: Investigation of the Effects of Motor Imagery to Facilitate Sensorimotor Re-Learning Training on Performance and Heart Rate Variability in Adolescent Basketball Players
Brief Title: Effects of Motor Imagery Training on Performance and Heart Rate Variability in Adolescent Basketball Players
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Emre Uysal, Lecturer, Ege University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-1251
Record Dates: First submitted 2023-05-23; First posted 2023-06-02 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2023-05

CONDITIONS: Motor Imagery
Keywords: Imagery; Exercise; Adolescent Basketball Players
MeSH Terms: conditions — Motor Activity | interventions — Control Groups

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): In addition to routine basketball technical-tactical training, the athletes in the experimental group will be given motor imagery training to facilitate sensorimotor relearning.
  Interventions: Other: Motor Imagery to Facilitate Sensorimotor Re-Learning Training
- Control Group (Active Comparator): Individuals in the control group will only continue their routine basketball technical-tactical training.
  Interventions: Other: Control Group

INTERVENTIONS:
Other: Motor Imagery to Facilitate Sensorimotor Re-Learning Training — In order to motor imagery to facilitate sensorimotor re-learning training will be given for 20 minutes a day, 3 days a week, for a total of 8 weeks. Basketball-specific movement patterns will be used (squat, single leg jump, side stepping, standing on one leg, squat on one leg, etc.). Exercises will be started from easy and progressed to more advanced levels. During the exercise, the person will not only be physically active, but will be asked to dynamically visualize the determined scenario. Thus, a holistic exercise program will be applied both physically and psychologically.
  Arms: Experimental Group
Other: Control Group — They will only continue their routine basketball technical-tactical training.
  Arms: Control Group

SUMMARY:
The aim of this study is to examine the investigation of the effects of motor imagery to facilitate sensorimotor re-learning training on performance and heart rate variability in adolescent basketball players.

DETAILED DESCRIPTION:
Motor imagery is defined as the mental process of simulating a certain action without any movement. In one study, researchers showed that motor imagery training activates the sensorimotor system and that brain plasticity resulting from actual movement execution also occurs as a result of motor imagery. When the literature is examined, it has been reported in studies that muscle strength may increase as a result of imagery training. However, there are also studies reporting that imagery training is effective on performance in basketball players.

Dynamic motor imagery, on the other hand, is a type of motor imagery in which the athletes adopt a harmonious body position and embody the spatial and/or temporal invariants of the movement without fully realizing it. According to a study, dynamic imagery training has a positive effect on free throw performance in basketball players. To facilitate sensorimotor relearning, which is a new training model, motor imagery training is an approach that approaches athletes with a holistic perspective, combining both physical exercises and dynamic motor imagery training. In a study, it was reported that training is more fun than just physical exercises . When the literature is examined; no study has been found examining the effects of motor imagery training on performance and heart rate changes in order to facilitate sensorimotor relearning in adolescent basketball players.

ELIGIBILITY:
Inclusion Criteria:

1. Being between the ages of 11-19
2. Playing licensed basketball for at least 2 years
3. Being a man

Exclusion Criteria:

1. Coming to the hospital with a musculoskeletal injury in the last 3 months
2. Not being willing to participate in the study

Ages: 11 Years to 19 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Balance | change from baseline at 8 weeks
  The balance of the athletes will be evaluated with the Y balance test.

SECONDARY OUTCOMES:
Muscle Power | change from baseline at 8 weeks
  The muscular power of the athletes will be evaluated with the vertical jump test.
Muscle Strength | change from baseline at 8 weeks
  The muscular strength of the athletes will be evaluated with a hand-held dynamometer. In this context, it will be done separately for the quadriceps femoris, hamstring and gastracnemius muscle groups.
Shooting Performance | change from baseline at 8 weeks
  Shooting performance of the athletes will be evaluated with the free throw test. Athletes shall attempt 10 free throws as successfully as possible. The researcher will hand the ball to the players before each shot. The number of successful free throws will be recorded from 0 to 10
Agility | change from baseline at 8 weeks
  The agility of the athletes will be evaluated with the hexagonal agility test. The test will be started while the athlete is standing on the tape strip placed in the middle of the hexagon marking the starting position. The researcher will start the stopwatch after giving the command "Ready, start" to the athlete. Each athlete will jump from the center of the hexagon to the outside of the hexagon with both legs. In this way, the athlete will turn around the hexagon 3 times and return to the center. The stopwatch will be stopped when the athlete returns to the center mark after 3 laps around the hexagon.
Heart Rate Variability | change from baseline at 8 weeks
  The heart rate variability will be performed with a heart rate monitor (Polar H10).

CONTACTS AND LOCATIONS:
Locations (1):
- Ege University, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided